CLINICAL TRIAL: NCT02732353
Title: Absorption and Muscle-stimulating Effect of Hydrolyzed and Minced Beef
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasper Dideriksen (Other)
Responsible Party: Sponsor-Investigator, Kasper Dideriksen, PhD, Post doc, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: H-15012327
Record Dates: First submitted 2016-03-30; First posted 2016-04-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Meat Protein Supplements; Protein Absorption and Amino Acid Availability; Muscle Protein Synthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minced beef (Active Comparator): Minced beef
  Interventions: Dietary Supplement: Minced beef
- Hydrolyzed beef (Experimental): Hydrolyzed beef
  Interventions: Dietary Supplement: Hydrolyzed beef

INTERVENTIONS:
Dietary Supplement: Minced beef — Cow meat protein supplement
  Arms: Minced beef
Dietary Supplement: Hydrolyzed beef — Cow meat protein supplement
  Arms: Hydrolyzed beef

SUMMARY:
To measure the absorption kinetics and postprandial amino acid availability after ingestion of minced beef compared with hydrolyzed beef in young males. Moreover, the basal muscle protein synthesis and the postprandial muscle protein synthetic response to minced beef and hydrolyzed beef ingestion are measured in young males. The postprandial muscle protein synthetic response is measured and compared during the early postprandial period (0-3 hours) after ingestion of the two meat products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-obese (BMI<30)

Exclusion Criteria:

* Chronic medical disease
* >5 hour of exercise weekly, except light activities such as stretching/gymnastics and bike-riding/walking as transportation

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change in skeletal muscle protein fractional synthetic rate | During the postprandial period (0-3 hrs).
  The fractional synthetic rate of skeletal muscle proteins (%/h) measured during the overnight fasted state and the postprandial state.

SECONDARY OUTCOMES:
Protein absorption | During the postprandial period (0-3 hrs).
  The change in venous plasma ring-2H5-phenylalanine enrichment after ingestion of meat protein, reflects the protein absorption from the meat protein products.
Plasma amino acid concentration | During the postprandial period (0-3 hrs).
  Change in venous plasma amino acid concentration after ingestion of meat protein.

CONTACTS AND LOCATIONS:
Overall Officials: Kasper Dideriksen, PhD, Principal Investigator — Bispebjerg Hospital; Lars Holm, PhD, Principal Investigator — Bispebjerg Hospital; Søren Reitelseder, PhD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No